CLINICAL TRIAL: NCT00831415
Title: A 10-Month Open-Label Evaluation Of The Long-Term Safety Of Desvenlafaxine Succinate Sustained Release In Japanese Adults With Major Depressive Disorder
Brief Title: Study Evaluating Long-Term Safety of Desvenlafaxine Succinate Sustained Release With Japanese Adult Subjects in Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-3350; B2061002
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Disorder
Keywords: Open-label Long-term extension study
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): DVS SR
  Interventions: Drug: desvenlafaxine succinate sustained release tablets

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained release tablets — 25-mg or 50-mg DVS SR tablets taken orally, once daily, at the same time each day. 100 mg dose will be supplied as 2 tablets of 50-mg tablet.
  Other Names: DVS-233; Pristiq

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of desvenlafaxine succinate sustained release tablets during 10-month open-label treatment of Japanese subjects with major depressive disorder (MDD).

The secondary objective is to evaluate the long-term response of subjects receiving desvenlafaxine succinate sustained release tablets by clinical global evaluation, general well-being and absence of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed double-blind therapy in short-term study for the indication of major depressive disorder (MDD), including scheduled evaluations, with no major protocol violations and no study events that, in the opinion of the investigator, would preclude the subject's entry into the long-term, open-label study.

Exclusion Criteria:

* Clinically important abnormalities on baseline (day 56 of the short-term study) physical examination, or any unresolved clinically significant abnormalities on electrocardiogram (ECG), laboratory test results, or vital signs recorded before day 56 in the previous short-term study for the indication of MDD.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Japan (17):
  - Pfizer Investigational Site, Aichi
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Fukushima
  - Pfizer Investigational Site, Gunma
  - Pfizer Investigational Site, Hiroshima
  - Pfizer Investigational Site, Hokkaido
  - Pfizer Investigational Site, Hyōgo
  - Pfizer Investigational Site, Ishikawa
  - Pfizer Investigational Site, Kanagawa
  - Pfizer Investigational Site, Kumamoto
  - Pfizer Investigational Site, Kyoto
  - Pfizer Investigational Site, Osaka
  - Pfizer Investigational Site, Saga
  - Pfizer Investigational Site, Saitama
  - Pfizer Investigational Site, Shiga
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-3350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 10-month, open-label, multicenter study of Japanese participants with Major Depressive Disorder (MDD) conducted from March 2009 to March 2011 at 61 sites in Japan.
Pre-assignment Details: A total of 304 participants who completed the short-term Core Study (NCT00798707 [3151A1-3359 / B2061003]) consented to enroll in this long-term, open-label, flexible dosing Extension study (NCT00831415 [3151A1-3350 / B2061002]). Baseline in this Extension study = Day 56 of the Core study.
Groups:
- DVS SR: Desvenlafaxine succinate sustained release formulation (DVS SR) flexible dose 25 milligrams per day (mg/day) up to 100 mg/day.
Period: Overall Study
Arm/Group | DVS SR
Started | 304
Completers for "Exposure" | 227 (Participants with ≥ 301 days of exposure to study drug and completed study day 308 evaluations.)
Study "Completers" | 227 (Defined as participants whose conclusion of study participation status was "study completed.")
Completed | 229 (In addition to Completers for Study includes 2 participants who discontinued after on-therapy period)
Not Completed | 75
Not completed — Adverse Event | 14
Not completed — Failed to return | 3
Not completed — Physician Decision | 6
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 35
Not completed — Unsatisfactory response - Efficacy | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- DVS SR: DVS SR flexible dose 25 mg/day up to 100 mg/day.
Arm/Group | DVS SR
Number analyzed (Participants) | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.45 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 155
Hamilton Psychiatric Scale for Depression-17 Item (HAM-D17) score [Mean (Standard Deviation); unit: scores on a scale] — HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4) with 0=none/absent and 4=most severe, for a maximum total score of 50. Higher scores indicate greater severity.
  scores on a scale | 12.86 (6.30)
Categorical scores on Clinical Global Impression-Improvement [CGI-I] [Number; unit: participants] — CGI-I is a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected. Baseline for CGI-I in this Extension study (NCT00831415 [3151A1-3350 / B2061002]) was measured against CGI-I baseline (Day -1) data in Core study (NCT00798707 [3151A1-3359 / B2061003]).
  participants
    1=Very much improved | 75
    2=Much improved | 81
    3=Minimally improved | 94
    4=No change | 51
    5=Minimally worse | 3
Clinical Global Impression-Severity of Illness [CGI-S] score [Mean (Standard Deviation); unit: scores on a scale] — CGI-S is a 7-point clinician rated scale to assess severity of current illness state. Range is 1 (normal - not ill at all) to 7 (among the most extremely ill). Higher score = more affected.
  scores on a scale | 3.25 (1.11)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Psychiatric Scale for Depression-17 Item (HAM-D17) Score
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4) with 0=none/absent and 4=most severe, for a maximum total score of 50. Higher scores indicate greater severity. FOT evaluation is defined as the last "on-therapy" evaluation, regardless of the number of days on therapy. Analysis on Observed cases (non-missing data) and Last observation carried forward (LOCF); LOCF method of imputation for any missing value at any visit.
Time Frame: Baseline (Extension Study) up to Day 308 or Final On-Therapy (FOT) Evaluation
Population: Intent to treat (ITT): all enrolled participants who received at least 1 dose of study treatment in Extension Study and at least 1 available post-baseline evaluation for any endpoint; (n)=number of participants with analyzable data at observation.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | DVS SR
Number analyzed (Participants) | 304
scores on a scale
  LOCF - change at FOT (n=304) | -4.76 [-5.47 to -4.05]
  Observed cases - change at Day 308 (n=224) | -5.82 [-6.61 to -5.03]

2. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression-Improvement (CGI-I)
Description: CGI-I is a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Day 308 or FOT Evaluation
Population: ITT; LOCF. Improvement measured against CGI-I baseline (Day -1) data in Core study (NCT00798707 [3151A1-3359 / B2061003]).
Measure: Number; unit: participants
Arm/Group | DVS SR
Number analyzed (Participants) | 304
participants
  1=Very much improved | 164
  2=Much improved | 82
  3=Minimally improved | 36
  4=No change | 15
  5=Minimally worse | 6
  6=Much worse | 1
  7=Very much worse | 0

3. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness [CGI-S] Score
Description: CGI-S is a 7-point clinician rated scale to assess severity of current illness state. Range is 1 (normal - not ill at all) to 7 (among the most extremely ill). Higher score = more affected.
Time Frame: Baseline (Extension Study) up to Day 308 or FOT Evaluation
Population: ITT; LOCF and Observed cases (non-missing data); (n)=number of participants with analyzable data at observation.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | DVS SR
Number analyzed (Participants) | 304
scores on a scale
  LOCF - change at FOT (n=304) | -0.82 [-0.94 to -0.70]
  Observed cases - change at Day 308 (n=224) | -0.95 [-1.09 to -0.80]

4. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study treatment was considered an AE without regard to possibility of causal relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be an SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly.
Time Frame: Baseline (Extension Study) up to Day 329 or 15 days after last dose of study treatment
Population: Safety population: all enrolled participants who received at least 1 dose of study treatment in this extension study.
Measure: Number; unit: percentage of participants
Arm/Group | DVS SR
Number analyzed (Participants) | 304
percentage of participants
  Adverse Events | 81.3
  Serious Adverse Events | 2.6

ADVERSE EVENTS:
Time Frame: Events were collected from the time of the signing of the informed consent form up to 15 days after the last dose of study treatment was administered.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | DVS SR
Serious Adverse Events (participants affected / at risk) | 8/304
Other Adverse Events (participants affected / at risk) | 247/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR (N=304)
Gastroenteritis (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Completed suicide (Psychiatric disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR (N=304)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 6
Ventricular extrasystoles (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 2
Motion sickness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 12
Vertigo (Ear and labyrinth disorders) | 5
Blepharospasm (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 10
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain lower (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 20
Aphthous stomatitis (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 17
Dental caries (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 29
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 3
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 3
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 6
Gastrointestinal disorder (Gastrointestinal disorders) | 3
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 38
Oral discomfort (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Chills (General disorders) | 2
Condition aggravated (General disorders) | 1
Device dislocation (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 7
Eye complication associated with device (General disorders) | 1
Fatigue (General disorders) | 4
Feeling abnormal (General disorders) | 6
Feeling hot (General disorders) | 1
Hangover (General disorders) | 1
Irritability (General disorders) | 3
Malaise (General disorders) | 8
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 4
Thirst (General disorders) | 10
Gallbladder polyp (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Allergy to arthropod sting (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Acute sinusitis (Infections and infestations) | 1
Adenoviral conjunctivitis (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 9
Gastroenteritis viral (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Herpangina (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 2
Influenza (Infections and infestations) | 7
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 122
Oral herpes (Infections and infestations) | 3
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Parotitis (Infections and infestations) | 1
Periodontal infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 2
Tinea infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Bone fissure (Injury, poisoning and procedural complications) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 9
Excoriation (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 2
Heat stroke (Injury, poisoning and procedural complications) | 1
Injury corneal (Injury, poisoning and procedural complications) | 2
Intentional overdose (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 4
Laceration (Injury, poisoning and procedural complications) | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Whiplash injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood potassium decreased (Investigations) | 1
Blood pressure diastolic increased (Investigations) | 1
Blood pressure increased (Investigations) | 6
Blood prolactin increased (Investigations) | 7
Blood triglycerides increased (Investigations) | 7
Blood uric acid increased (Investigations) | 4
Blood urine present (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 8
Glucose urine present (Investigations) | 2
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Lipids abnormal (Investigations) | 1
Lipids increased (Investigations) | 1
Liver function test abnormal (Investigations) | 6
Neutrophil count decreased (Investigations) | 1
Occult blood positive (Investigations) | 1
Platelet count decreased (Investigations) | 1
Protein urine present (Investigations) | 3
Red blood cell count decreased (Investigations) | 2
Urine ketone body present (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 19
White blood cell count decreased (Investigations) | 3
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperphagia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 17
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 3
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 36
Dizziness postural (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 36
Hypoaesthesia (Nervous system disorders) | 6
Intercostal neuralgia (Nervous system disorders) | 1
Irregular sleep phase (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 38
Tremor (Nervous system disorders) | 3
Visual field defect (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Anger (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 14
Depression suicidal (Psychiatric disorders) | 3
Dissociative disorder (Psychiatric disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Impulsive behaviour (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 13
Insomnia related to another mental condition (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 2
Nervousness (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Self injurious behaviour (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 12
Withdrawal syndrome (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Endometriosis (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2
Genital haemorrhage (Reproductive system and breast disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Menstruation delayed (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 5
Metrorrhagia (Reproductive system and breast disorders) | 2
Oligomenorrhoea (Reproductive system and breast disorders) | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 1
Sexual dysfunction (Reproductive system and breast disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 5
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Urticaria thermal (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1
Pregnancy of partner (Social circumstances) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.